CLINICAL TRIAL: NCT00952965
Title: Clinical Testing Report for Wrist-used Electronic Blood Pressure Monitor
Brief Title: Wrist-used Blood Pressure Monitor Clinical Test (Cuff Range: 14cm-25cm)
Acronym: WBPMCT
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Liu Yi, Andon Health co., LTD
Other Study IDs: AndonHealth2
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Blood Pressure
Keywords: BP

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- blood pressure monitor: wrist circumference: 14cm-25cm
- stethoscopy: wrist circumference: 14cm-25cm

SUMMARY:
The purpose of this study is to monitor the blood pressure level of the patient using a wrist cuff ranged 14 cm-25 cm.

ELIGIBILITY:
Inclusion Criteria:

* wrist circumference: 14 cm-25 cm

Exclusion Criteria:

* none

Ages: 23 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: resident of a community.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
level of blood pressure | 10 s

CONTACTS AND LOCATIONS:
Overall Officials: Qi Sun, Principal Investigator — Andon Health Co., Ltd
Locations (1):
- Beichen hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Wong SN, Tz Sung RY, Leung LC. Validation of three oscillometric blood pressure devices against auscultatory mercury sphygmomanometer in children. Blood Press Monit. 2006 Oct;11(5):281-91. doi: 10.1097/01.mbp.0000209082.09623.b4. PMID 16932037